CLINICAL TRIAL: NCT05016310
Title: A Randomized, Open-label Study of High-Dose Vitamin D Versus Standard of Care Vitamin D Supplementation to Evaluate the Impact on Bone Health in Young Women With Early Stage Breast Cancer
Brief Title: A Study of High-Dose Vit D Versus Standard of Care Vit D Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCI-BRE-VITD-001; 00055909 (Other: Advarra IRB); LCI-BRE-VITD-001 (Other: LCI)
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Breast; Breast Cancer; Osteoporosis
Keywords: Bone Density
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Vit D (Experimental): High Dose Vitamin D
  Interventions: Dietary Supplement: High Dose Vitamin D
- SOC Vit D (Active Comparator): Standard of Care Vitamin D
  Interventions: Dietary Supplement: Standard of Care Vitamin D

INTERVENTIONS:
Dietary Supplement: High Dose Vitamin D — High dose vitamin D: Subjects will receive 50,000 IU vitamin D2 weekly x 16 weeks followed by 4,000 IU of vitamin D3 daily with a goal 25(OH)D level of ≥45 but ≤80 ng/mL.
  Arms: High Vit D
Dietary Supplement: Standard of Care Vitamin D — Standard of Care Vitamin D: Vitamin D will be supplemented to 25(OH)D levels, with a goal 25(OH)D level of >30 ng/mL according to Endocrine Society Practice Guidelines.
  Arms: SOC Vit D

SUMMARY:
This is a randomized study evaluating the effects of early intensive vitamin D supplementation compared to standard of care vitamin D supplementation on bone health over an 18 month period.

DETAILED DESCRIPTION:
This is a randomized, open-label study designed to evaluate the effect of high dose vitamin D versus standard of care vitamin D supplementation on bone health and arthralgias. The randomization will be stratified by hormone receptor status (positive versus negative). The primary objective is to compare the effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on bone health, as measured by percent change from baseline in bone mineral density (g/cm2), in young women with non-metastatic breast cancer who receive systemic therapy.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age; 45 years at the time of consent
3. Female
4. Histological or cytological confirmation of breast cancer clinical or pathologic stages 0-III
5. Patient has been recommended to initiate systemic therapy for breast cancer. It is preferable for patient to enroll prior to systemic therapy initiation. However, enrollment will be allowed if systemic therapy has been initiated within 4 weeks prior to enrollment (randomization).

   Note: Patients who undergo only surgery and/or radiotherapy alone would not qualify for the study.
6. Systemic therapy for breast cancer is planned
7. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study
8. Previous vitamin D supplementation allowed, as long as patient is agreeable to stop previous dosing at the time of trial enrollment, to comply with trial procedures including a baseline 25(OH)D level, and is otherwise determined to be appropriate for enrollment

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

1. Uncontrolled intercurrent illness/medical condition or psychiatric illness/social situations that would limit compliance with study requirements as determined by the Investigator
2. Patients will undergo breast surgery and/or radiotherapy alone without planned neoadjuvant and/or adjuvant anti-cancer drug therapy.
3. Baseline 25(OH)D level <10ng/mL or >80ng/mL
4. Baseline serum corrected calcium level of >10.3mg/dL
5. Bone mineral density less than the expected range for age on baseline DEXA scan (defined as Z-score </= -2.0)
6. Breast cancer with distant metastasis
7. History of previous breast cancer
8. Postmenopausal, as confirmed by the lack of menses >/=12 months and/or ovarian function laboratories (estradiol, FSH) consistent with menopause (if any of two values outside of menopausal range and subject had menses within 12 months, subject would be considered perimenopausal or premenopausal and therefore eligible for enrollment)
9. Pregnancy or lactation
10. History of bone disease, including Paget's bone disease or osteomalacia
11. Concurrent rheumatoid or other inflammatory arthritis
12. Concurrent or prior treatment with bisphosphonates
13. Use of oral corticosteroids within the last 30 days prior to randomization
14. Concurrent treatment for thyroid deficiency
15. BMI <18.5
16. Currently receiving treatment for tuberculosis, or planning to receive treatment for tuberculosis during breast cancer treatments
17. History of another primary cancer that required systemic treatment within the last 5 years
18. Any of the following kidney diseases at the time of randomization: active chronic kidney disease >/= stage 3, history of kidney stones, sarcoidosis
19. Gastrointestinal disease that would limit the absorption of pill therapy (i.e. celiac disease, gastric bypass surgery)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in bone mineral density (g/cm^2) from baseline to the Year 1 DEXA scan | 15 months (12 plus a +3 month calendar window)
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on bone health, as measured by percent change from baseline in bone mineral density (g/cm2) to the Year 1 planned DEXA scan, in young women with non-metastatic breast cancer who receive systemic therapy.

SECONDARY OUTCOMES:
25(OH) D level over time | 18 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm 25(OH) D levels in young women with non-metastatic breast cancer who receive systemic therapy.
PRAI questionnaire results over time | 18 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on PRAI questionnaire results in young women with non-metastatic breast cancer who receive systemic therapy.
Overall satisfaction with pain control over time | 18 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on overall satisfaction with pain control in young women with non-metastatic breast cancer who receive systemic therapy.
Skeletal complications over time | 18 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on skeletal complications in young women with non-metastatic breast cancer who receive systemic therapy.

OTHER OUTCOMES:
Vitamin D administration | 18 months
  Descriptively summarize vitamin D administration for the high dose vitamin D arm and for the current standard vitamin D treatment administration algorithm in young women with non-metastatic breast cancer who receive systemic therapy.
Adverse events of special interest | 19 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on adverse events of special interest (vitamin D related headaches, irritability, spasticity, nausea, vomiting, and hypercalcemia) in young women with non-metastatic breast cancer who receive systemic therapy.
Adverse events of special interest leading to vitamin D dose modifications or discontinuations | 18 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on adverse events of special interest (vitamin D related headaches, irritability, spasticity, nausea, vomiting, and hypercalcemia) that results in vitamin D dose modifications or discontinuations in young women with non-metastatic breast cancer who receive systemic therapy.
Serious adverse events | 19 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on serious adverse events in young women with non-metastatic breast cancer who receive systemic therapy.
Treatment discontinuation due to vitamin D non-compliance | 18 months
  Compare effect of high dose vitamin D to the current standard vitamin D treatment administration algorithm on treatment discontinuation due to vitamin D intake non-compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Heeke, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT05016310/ICF_000.pdf